CLINICAL TRIAL: NCT02980016
Title: A Randomised, Pragmatic, Open-Label Trial To Evaluate The Effect Of Three Months Of High Dose Rifapentine Plus Isoniazid Administered As A Single Round Or Given Annually In HIV-Positive Individuals
Brief Title: Evaluation of the Effect of 3HP vs Periodic 3HP vs 6H in HIV-Positive Individuals
Acronym: WHIP3TB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Aurum Institute (Other); London School of Hygiene and Tropical Medicine (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3HP-AUR1-1-170
Record Dates: First submitted 2016-11-21; First posted 2016-12-02 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3HP (rifapentine + isoniazid) (Active Comparator): Once weekly rifapentine (at a dose of 900 mg) plus isoniazid (at a dose of 900 mg), (with adjustment for participants weighing ≤50 kg) given for 12 weeks in Study Year 1
  Interventions: Drug: rifapentine + isoniazid
- p3HP (rifapentine + isoniazid) (Active Comparator): Once weekly rifapentine (at a dose of 900 mg) plus isoniazid (at a dose of 900 mg), (with adjustment for participants weighing ≤50 kg) given for 12 weeks in Study Years 1 and 2
  Interventions: Drug: rifapentine + isoniazid
- 6H (Active Comparator): Daily self-administered isoniazid (at a dose of 300 mg/daily) (with adjustment for participants weighing ≤24 kg) given for 26 weeks (6 months) in Study Year 1
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: rifapentine + isoniazid — Rifapentine + isoniazid Once weekly rifapentine (at a dose of 900 mg) plus isoniazid (at a dose of 900 mg), with adjustment for participants weighing ≤50 kg
  Other Names: Priftin (rifapentine)
  Arms: 3HP (rifapentine + isoniazid); p3HP (rifapentine + isoniazid)
Drug: Isoniazid — Daily self-administered isoniazid (at a dose of 300 mg/daily), with adjustment for participants weighing ≤24 kg
  Other Names: Winthrop (isoniazid)
  Arms: 6H

SUMMARY:
This study is a parallel, two part, open label, individually randomized, pragmatic trial among HIV-positive individuals. Part A compares a single round of weekly high dose rifapentine plus isoniazid for three months (3HP) to six months of daily isoniazid (6H). Part B compares periodic 3HP (p3HP) to a single round of 3HP.

DETAILED DESCRIPTION:
Part A: A randomised controlled trial of 3HP vs 6H [enrollment starts concurrently with Part B]

Justification: The World Health Organization (WHO) recommends at least six months of isoniazid (6H) for persons living with HIV. However, 6H remains poorly implemented in most high burden tuberculosis (TB) countries. In its 2015 guidelines, WHO includes 3HP as an latent tuberculosis infection (LTBI) treatment option for high-income and upper middle-income countries with TB incidence rates <100/100,000. One trial comparing 3HP to 6H in a high burden country suggests that a single round of 3HP has less toxicity, better treatment completion rates, and similar efficacy in preventing TB. The purpose of comparing a single round of 3HP to 6H is to demonstrate the feasibility of implementing 3HP in high burden countries, to explore its safety and effectiveness, and to generate evidence to guide a WHO recommendation for the use of 3HP in high burden settings.

Sample size: If we assume 85% of patients in the 6H arm complete treatment as defined above, with 400 patients in the 6H arm and 3600 patients in the 3HP arm we will have 82% power to detect an increase in treatment completion of 5% (To -90%) in the 3HP arm. If treatment completion in the 6H arm is 75%, we will have approximately 90% power to detect an increase in treatment completion of 7% in the 3HP arm.

Analysis: Treatment completion will be compared by study arm using Fishers Exact test, and associated risk difference and 95% confidence interval (CI).

Part B: A randomised controlled trial of 3HP vs p3HP [enrollment starts concurrently with Part A]

Justification: A single round of 3HP has been shown to be non-inferior to 9 months of isoniazid (9H) in persons at high risk of developing TB in low and middle TB burden settings. Similarly, a single round of 3HP has demonstrated similar efficacy in preventing active TB when compared to 6H among HIV-positive, tuberculin skin test (TST)-positive adults in the high burden setting of South Africa. In high burden settings, 6H and 3HP provide protection of limited duration probably due to high ongoing transmission and reinfection. Continuous isoniazid preventive therapy has been shown to provide more durable protection in high burden settings, but is not currently policy outside of a handful of countries, and the actual uptake is poor. Giving 3HP periodically may provide durable protection, be easier for health systems to implement, and may be associated with better adherence and fewer side effects.

Sample size: Assuming a cumulative TB incidence of 5% over 2 years in the control (3HP) arm, an overall loss to follow-up of 10% by year 2, a two-sided type I error of 5%, 1:1 randomisation, a superiority comparison and 1800 participants per arm, we have 80% power to detect a 40% reduction in cumulative TB incidence from months 0 to 24.

Analysis: The analysis will compare 3HP and p3HP with two years of follow up. Cumulative TB incidence will be determined by combining incident TB cases identified over the 24 months of follow up AND prevalent TB cases identified at the 12 and 24 month culture survey. Data will be reported as a risk difference and odds ratio and their associated 95% CIs, adjusting for randomisation strata. The secondary outcome comparing the effectiveness of p3HP to 3HP from month 13 to 24 (during which time the greatest effect is likely to be evident) will be conducting using the same analytic methods. The results of Part B will be disseminated subsequent to the results of Part A.

ELIGIBILITY:
Inclusion Criteria:

* At least two years of age
* Known HIV infection
* Antiretroviral therapy (ART) ineligible or on ART for ≥3 months

Exclusion Criteria:

* Confirmed or suspected TB disease
* Likely to move from the study area during the study period
* Known exposure to TB cases with known or suspected resistance to isoniazid or rifampicin in the source case
* TB treatment within the past year
* TB preventive therapy within the last year
* Sensitivity or intolerance to isoniazid or rifamycins
* Suspected acute hepatitis or known chronic liver disease
* ALT/AST >5 times the upper limit of normal (regardless of symptoms of hepatitis)
* Pregnancy or breastfeeding
* Women of childbearing potential who are unable or unwilling to use contraception
* Self-reported alcohol use exceeding 28 units per week for men, or 21 units for women

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4027 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Treatment completion (part A) | 1 year
  Number of participants without evidence of active TB at enrollment who complete treatment, defined as:
  Proportion of participants in 3HP group self-reporting treatment completion of ≥11 doses in a 16-week period
  ; Proportion or participants in 6H group self-reporting treatment completion of ≥167 doses over an 34 week (8-month) period
TB incidence (part B) | 2 years
  Number of participants without evidence of active TB at enrollment who are diagnosed with active TB meeting the definition: Confirmed tuberculosis: Culture-positive, Xpert MTB/RIF-positive, or smear-positive for M. tuberculosis from any site in adults and children OR Clinical tuberculosis: Started on treatment for TB in adults and children

SECONDARY OUTCOMES:
TB incidence (part A) | 1 year
  Number of participants without evidence of active TB at enrollment who are diagnosed with active TB meeting the definition: Confirmed tuberculosis: Culture-positive, Xpert MTB/RIF-positive, or smear-positive for M. tuberculosis from any site in adults and children OR Clinical tuberculosis: Started on treatment for TB in adults and children
All-cause mortality (part A) | 1 year
  Number of participants without evidence of active TB at enrollment who die from any cause
Permanent discontinuation of therapy due to treatment-related adverse events (part A) | 1 year
  Number of participants without evidence of active TB at enrollment who permanently discontinue therapy due to an adverse drug reaction
TB incidence (part B) | 1 year
  Number of participants without evidence of active TB during enrollment who are diagnosed with active TB meeting during the second year of follow-up. The definition of active TB is: Confirmed tuberculosis: Culture-positive, Xpert MTB/RIF-positive, or smear-positive for M. tuberculosis from any site in adults and children OR Clinical tuberculosis: Started on treatment for TB in adults and children
Treatment completion (part B) | 2 years
  Number of participants without evidence of active TB at enrollment who complete treatment, defined as: Proportion of participants in 3HP group self-reporting treatment completion of ≥11 doses in a 16-week period; Proportion or participants in p3HP group self-reporting treatment completion of ≥22 doses over two annual 16-week periods
All-cause mortality (part B) | 2 years
  Number of participants without evidence of active TB at enrollment who die from any cause
Permanent discontinuation of therapy due to treatment-related adverse events (part B) | 2 years
  Number of participants without evidence of active TB at enrollment who permanently discontinue therapy due to an adverse drug reaction
Cost per TB case prevented | 2 years
  Cost per TB case prevented
Cost per death averted | 2 years
  Cost per death averted
Cost per disability adjusted life year (DALY) averted by study arm | 2 years
  Cost per disability adjusted life year (DALY) averted by study arm

OTHER OUTCOMES:
IGRA conversions (part A) | 1 year
  Number of IGRA-negative participants without evidence of active TB at enrollment with the occurrence of IGRA conversions at the end of year 1
IGRA reversions (part A) | 1 year
  Number of IGRA-positive participants without evidence of active TB at enrollment with the occurrence of IGRA reversions at the end of year 1
Incidence of TB resistant to isoniazid and/or rifapentine | 2 years
  Number of individuals without evidence of active TB at enrollment who are diagnosed with active TB resistant to isoniazid and/or rifapentine

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, MBBCh, PhD, Principal Investigator — Aurum Institute
Locations (1):
- The Aurum Institute NPC, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Sterling TR, Moro RN, Borisov AS, Phillips E, Shepherd G, Adkinson NF, Weis S, Ho C, Villarino ME; Tuberculosis Trials Consortium. Flu-like and Other Systemic Drug Reactions Among Persons Receiving Weekly Rifapentine Plus Isoniazid or Daily Isoniazid for Treatment of Latent Tuberculosis Infection in the PREVENT Tuberculosis Study. Clin Infect Dis. 2015 Aug 15;61(4):527-35. doi: 10.1093/cid/civ323. Epub 2015 Apr 22. PMID 25904367
- [Background] Sterling TR, Benson CA, Shang N. Tolerability among HIV-infected persons of three months of once-weekly rifapentine + INH (3HP) vs. 9 months of daily INH (9H) for treatment of latent tuberculosis infection. In: International AIDS Society Conference. Washington, DC.; 2012.
- [Background] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833
- [Background] Villarino ME, Scott NA, Weis SE, Weiner M, Conde MB, Jones B, Nachman S, Oliveira R, Moro RN, Shang N, Goldberg SV, Sterling TR; International Maternal Pediatric and Adolescents AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Treatment for preventing tuberculosis in children and adolescents: a randomized clinical trial of a 3-month, 12-dose regimen of a combination of rifapentine and isoniazid. JAMA Pediatr. 2015 Mar;169(3):247-55. doi: 10.1001/jamapediatrics.2014.3158. PMID 25580725
- [Derived] Churchyard G, Cardenas V, Chihota V, Mngadi K, Sebe M, Brumskine W, Martinson N, Yimer G, Wang SH, Garcia-Basteiro AL, Nguenha D, Masilela L, Waggie Z, van den Hof S, Charalambous S, Cobelens F, Chaisson RE, Grant AD, Fielding KL; WHIP3TB Study Team. Annual Tuberculosis Preventive Therapy for Persons With HIV Infection : A Randomized Trial. Ann Intern Med. 2021 Oct;174(10):1367-1376. doi: 10.7326/M20-7577. Epub 2021 Aug 24. PMID 34424730